CLINICAL TRIAL: NCT00317512
Title: A Multi-Center,Randomized,Double-Blind,Placebo-Controlled,Dose Finding Pilot Study, to Evaluate Safety/Feasibility of HBOC-201 in Elective Percutaneous Coronary Revascularization of Subjects With Acute Coronary Syndromes
Brief Title: Pilot Study of Hemoglobin Based Oxygen Therapeutics in Elective Coronary Revascularization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biopure Corporation (Industry)
Responsible Party: Biopure Corporation, Biopure Corporation
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: COR-0001
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Angina Pectoris; Unstable Angina; Myocardial Infarction
Keywords: Hemoglobin Based Oxygen carrier; HBOC 201; Percutaneous Revascularization; Percutaneous Coronary Intervention; Non ST-segment Elevation Myocardial Infarction; Tissue Oxygenation; Transluminal Percutaneous Coronary Angioplasty
MeSH Terms: conditions — Angina Pectoris; Angina, Unstable; Myocardial Infarction | interventions — Percutaneous Coronary Intervention; HBOC 201; HES 130-0.4

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Voluven will be administered at 7.7 ml/min over 15 minutes,followed by Voluven at 7.7 ml/min over 15 minutes
  Interventions: Procedure: Percutaneous Coronary Revascularization; Drug: Voluven
- 2 (Active Comparator): HBOC-201 will be administered at 7.7 ml/min over 15 minutes,followed by Voluven at 7.7 ml/min over 15 minutes
  Interventions: Procedure: Percutaneous Coronary Revascularization; Drug: Hemoglobin-Based Oxygen Carrier-201 (HBOC-201); Drug: Voluven
- 3 (Experimental): HBOC-201 will be administered at 7.7 ml/min over 15 minutes,followed by HBOC-201 at 7.7 ml/min over 15 minutes
  Interventions: Procedure: Percutaneous Coronary Revascularization; Drug: Hemoglobin-Based Oxygen Carrier-201 (HBOC-201)

INTERVENTIONS:
Procedure: Percutaneous Coronary Revascularization
Drug: Hemoglobin-Based Oxygen Carrier-201 (HBOC-201)
  Arms: 2; 3
Drug: Voluven
  Arms: 1; 2

SUMMARY:
The purpose of this study is to assess the safety and feasibility of a novel oxygen carrying solution, HBOC-201, in the setting of PCI for Acute Coronary Syndromes from randomization til hospital discharge.

DETAILED DESCRIPTION:
Acute coronary syndromes are due to an acute or subacute primary reduction of myocardial oxygen supply provoked by disruption of an atherosclerotic plaque associated with inflammation, thrombosis, vasoconstriction and microembolization. Occlusive thrombosis superimposed on a ruptured atheroma in an epicardial coronary artery is firmly established as the immediate cause of an acute ST-segment Elevation Myocardial Infarction (STEMI). Rapid restoration of blood flow (oxygen supply) to jeopardized myocardium limits necrosis and reduces mortality. This can be accomplished medically with a thrombolytic agent, or mechanically, with so-called primary balloon angioplasty or stenting. Primary percutaneous coronary intervention (PCI) has become the preferred therapy for STEMI in most developed countries.

HBOC-201 is a solution belonging to a new class of biologic oxygen therapeutics, hemoglobin based oxygen carriers. HBOC-201 is a crosslinked and glutaraldehyde-polymerized hemoglobin (Hb) extracted from isolated bovine red blood cells. On a gram-for-gram basis, HBOC-201 was calculated to be approximately three times more potent than stored fresh red blood cell hemoglobin at restoring baseline tissue oxygenation following severe acute anemia. Evaluation of this Hemoglobin Based Oxygen Carrier has been undertaken in 57 preclinical studies and 21 human clinical trials. The compound is under review by the US FDA and has been approved in the Republic of South Africa. However, HBOC-201 has not yet been evaluated in the setting of this disease (narrowing of a coronary artery).

Biopure will be studying the safety and feasibility of HBOC-201 in patients with typical symptoms of Unstable Angina or Non ST-segment Elevation Myocardial Infarction eligible to undergo invasive revascularization through a PCI procedure.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided before initiation of any study-related procedure, and before any pre-procedural sedation, and agreement to comply with all protocol-specified procedures
* Acute Coronary Syndrome (Stable and unstable angina or non ST segment Elevation Myocardial Infarction (UA/non-STEMI) [Braunwald class I-III Class B], Appendix 1).
* Single vessel disease of the Left Coronary Artery (LCA)
* One vessel disease of the Right Coronary Artery (RCA)
* Have a single de novo lesion
* Older than 18 years and younger than 75 years of age
* Eligible to undergo PCI on the target vessel

Exclusion Criteria:

* Previous Q-wave myocardial infarction
* Congestive heart failure with Left ventricular Ejection Fraction <35%
* Confirmed pregnancy
* Anemia to a hemoglobin level <8.5g/dl
* Systemic mastocytosis
* History of known haemorrhagic stroke at any time or any stroke less than or equal to 30 days prior to randomization
* Severe hypertension (>180/110mmHG) not adequately controlled by antihypertensive therapy at time of study entry
* Need for mechanical ventilation
* Renal impairment: Creatinine > 1.6mg/dl
* Known history of COPD with FEV 1s < 1.0 liter
* Contra-indications to the use of adenosine, i.e.History of bronchospasm and/or ongoing therapy with theophylline derivatives, >1 degree atrioventricular block in the absence of a functioning electronic pacemaker and treatment with dipyridamole within the prior 24 hours
* Patients with significant hemodynamic compromise and/or cardiogenic shock requiring inotropic or pressor support or pulmonary edema
* History of or clinical documentation of severe aortic/mitral valve stenosis, significant aortic valve insufficiency
* Participation in another trial with an investigational drug or device (of other investigations) including the follow-up period, within the last 30 days before enrollment
* Inability or unwillingness to perform 30 day follow up
* Concomitant disease that interferes with prognosis (life expectancy of less than or equal to 6 months
* Contra-indications to standard drugs for coronary intervention and coronary heart disease: aspirin, heparin, low molecular weight heparin, clopidogrel, contrast dye
* Patient weight > 110kg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-12; Primary Completion 2005-04 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety
In hospital thrombotic events
Anaphylactic reactions
Inflammatory reactions
Substantial changes to systemic & coronary hemodynamics
Circulatory overload
Renal dysfunction
Untoward drug interaction effects
substantial changes in laboratory parameters
Life threatening cardiac arrhythmias
Other adverse events
Feasibility:
Number of subjects requiring premature discontinuation of study drug for clinical or logistical reasons

CONTACTS AND LOCATIONS:
Overall Officials: P W Serruys, Professor, Principal Investigator — University Medical Center Rotterdam
Locations (6):
- Belgium (2):
  - Site # 5 Onze Lieve Vrouw Ziekenhuis (OLVZ), Aalst
  - Site # 6 Antwerpen, Antwerp
- Site # 2 Herzzentrum, Leipzig, Germany
- Netherlands (3):
  - Site # 3 OLVG Amsterdam, Amsterdam
  - Site # 4 Academisch Medisch Centrum (AMC), Amsterdam
  - Site # 1 Erasmus Medical Center, Rotterdam

REFERENCES:
- [Result] Serruys PW, Vranckx P, Slagboom T, Regar E, Meliga E, de Winter RJ, Heyndrickx G, Schuler G, van Remortel EA, Dube GP, Symons J. Haemodynamic effects, safety, and tolerability of haemoglobin-based oxygen carrier-201 in patients undergoing PCI for CAD. EuroIntervention. 2008 Mar;3(5):600-9. doi: 10.4244/eijv3i5a108. PMID 19608488